CLINICAL TRIAL: NCT00301535
Title: Enhancement of Tissue Preservation During Cardiopulmonary Bypass With HBOC-201 (Registry Study)
Brief Title: A Study of Hemopure® to Enhance Tissue Preservation During Cardiopulmonary Bypass Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopure Corporation (Industry)
Responsible Party: Biopure, Biopure
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOEU003
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass Graft; memory loss after cardiac surgery; side effects of bypass
MeSH Terms: conditions — Coronary Artery Disease | interventions — HBOC 201

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: HBOC-201 (hemoglobin glutamer-250 bovine)
- 2 (No Intervention)

INTERVENTIONS:
Drug: HBOC-201 (hemoglobin glutamer-250 bovine) — HBOC-201 is an investigational solution of purified, glutaraldehyde-polymerized bovine hemoglobin with a concentration of hemoglobin of 13 ± 1 g/dL
  Arms: 1

SUMMARY:
The purpose of this study is to determine if Hemopure® will enhance tissue preservation during Cardiopulmonary Bypass surgery.

DETAILED DESCRIPTION:
The primary objective is to determine the safety and feasibility of administering Hemopure® (HBOC-201) to reduce myocardial necrosis, as measured by CK-MB enzyme elevation, and enhance tissue preservation during cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18 and 80.
* Subject is an acceptable candidate for CABG.
* Subject is scheduled for CABG (without planned valvular repair or replacement) by cardiopulmonary bypass.
* Subject signs informed consent
* Subject and the treating physician agree that subject can comply with all study procedures and follow-up visit at time of subject screening.

Exclusion Criteria:

* Pre-operative myocardial infarction, defined as CK-MB level > 2 times upper limit of normal 24 hours prior to CABG surgery.
* Renal failure defined as serum creatinine greater 220 µmol/L
* Subject has an ejection fraction ≤ 30% (as measured by Echocardiography within 30 days of study enrollment).
* Active infection.
* History of prior stroke within last six months or history of prior stroke with residual neurological deficit.
* Transient Ischemic attack within last 6 months.
* Subject has a history of coagulopathy.
* Subject is pregnant or currently breastfeeding.
* History of allergy to beef products.
* Pre-operative cardiogenic shock defined as cardiac index ≤ 1.8.L/min/m2 despite the use of vasopressors.
* Underlying medical conditions that would limit subject's life expectancy to less than 12 months.
* Severe pulmonary disease [based upon clinical diagnosis or pulmonary function tests (FEV <1 liter), if available] that may interfere with weaning subject from ventilator.
* History of acute central nervous disorder (e.g., seizure or traumatic injury).
* Severe hypertension (≥ 160/90 mm Hg) that cannot be medically controlled despite treatment with two antihypertensive therapies.
* Severe liver dysfunction as defined by total bilirubin ≥ 51 µmol/L or 2 times the site normal limit of AST or ALT activity.
* Subject has systemic mastocytosis.
* Subject has any condition that predisposes the subject to systemic mast cell degranulation or hypersensitivity reactions or a history of severe allergic reactions to drugs or environmental allergens.
* Subject has participated in another investigational drug, biologic or device study within 30 days prior to study enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-07 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Rate of peak CK-MB elevation ≥ 5X upper limit of normal | Baseline; Peri-op; Days 1,2,3 post procedure; Discharge or Day 6 post procedure(whichever is earlier)

SECONDARY OUTCOMES:
MACE @ discharge and 30 days post surgery; Change in renal function; Renal failure; Increased Cardiac Troponin T; Death rate; MI/stroke; Supplemental RBC transfusions; Total units RBC and HBOC-201; Intra Aortic Balloon Pump use, pump time; New onset CHF | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: A. Gerson Greenburg, MD, Ph.D, Study Director — Biopure Corporation
Locations (3):
- Thessaloniki Heart Institute - St. Luke's Hospital, Thessaloniki, Greece
- Milpark Hospital, Johannesburg, South Africa
- Oxford Heart Centre - John Radcliffe Hospital, Headington, Oxfordshire, United Kingdom